CLINICAL TRIAL: NCT02465970
Title: BRAINSTIM : Effects of Transcranial Direct Current Stimulation (TDCS) in Drug-resistant Partial Epilepsy
Brief Title: Effects of Transcranial Direct Current Stimulation (TDCS) in Drug-resistant Partial Epilepsy
Acronym: BRAINSTIM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 35RC14_9808
Record Dates: First submitted 2015-06-01; First posted 2015-06-09 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Epilepsy
Keywords: Transcranial Direct Current Stimulation
MeSH Terms: conditions — Epilepsy | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TDCS session (Experimental): Intervention : Stimulation is applied during a 60 min session with STARSTIM
  Interventions: Device: STARSTIM
- TDCS Placebo (Placebo Comparator): Intervention : Stimulation is not applied during a 60 min session with STARSTIM
  Interventions: Device: sham TDCS

INTERVENTIONS:
Device: STARSTIM — Multifocal transcranial direct current stimulation.
  * CE-marked device, comprising a cap with 2 to 8 electrodes, connected with a programmable mobile stimulator.
  * The stimulation is applied during a 60 min session
  Other Names: TDCS TransCranial Direct Current Stimulation
  Arms: TDCS session
Device: sham TDCS
  Arms: TDCS Placebo

SUMMARY:
Drug-resistant partial epilepsy has a heavy impact on quality of life and sometimes on life expectancy itself. Only a minority of patients may benefit from a curative epilepsy surgery. Neurostimulation, which can be an effective add-on treatment, is currently mainly represented by vagus nervus stimulation. Transcranial direct current stimulation, a non -invasive technique already used in other areas of neurology, may be efficient on some partial epilepsies, in particular through the individual configuration of stimulation, made possible by recent technological advances.

Main goal : To study the effect of transcranial electrical stimulation on the frequency of seizures in patients with drug-resistant partial epilepsy.

Hypothesis : Reduction of 50% or more in the frequency of occurrence of seizures within 24 hours following an individually configured TDCS session: responders in real TDCS vs placebo stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 15 years;
* Patients with drug-partial resistant epilepsy with the following characteristics:
* Disabling epilepsy despite an optimized pharmacological treatment.
* An average of one seizure a day or more during the week preceding the inclusion
* Focal epilepsy in which epileptogenic zone is documented by paraclinical examinations consistent with clinical data
* Existence of measurable EEG markers of epilepsy
* Anti-epileptic drug treatment unmodified during the 2 weeks preceding the inclusion no change to treatment planned during the study.
* Signed informed consent.

Exclusion Criteria:

* Patients under 15 years;
* Patients in which a standard quality EEG recording is not possible
* Patients with ictal bradycardia or ictal syncope ;
* Patients with heart disease which may result in heart arrhythmia ;
* Incapacitated patients (curatorship, guardianship), patients deprived of liberty.
* Pregnant or lactating women
* Vagus nervus stimulation is not an exclusion criteria

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Reduction of 50% or more in the frequency of occurrence of seizures within 24 hours following an individually configured TDCS session: responders in real TDCS vs placebo stimulation. | 24 hours

SECONDARY OUTCOMES:
Clinical : - Significant reduction of the frequency of occurrence of seizures within 24 hours, 48 hours, and 7 days following a session of TDCS. | 24 hours until 7 days
Clinical : - Reduction in the duration of seizures | 6 months
Electrophysiological : Decrease of epileptic EEG paroxysms at 8 and 24 hours after a TDCS session | 8-24 hours
- Clinical : If appropriate, reduction of the frequency of occurrence of secondary generalized seizures. | 6 months
-Clinical : Improvement in the quality of life within 7 days following a TDCS session | 7 days
Electrophysiological : - Decrease of epileptic EEG paroxysms immediately following a TDCS session. | up to 1 min

CONTACTS AND LOCATIONS:
Overall Officials: BIRABEN Arnaud, Principal Investigator — Rennes HU
Locations (1):
- Service de Neurologie, Rennes, France